CLINICAL TRIAL: NCT05435157
Title: Comparative Observational Study of Residual Gastric Volume Measured by Ultrasound After Preoperative Fasting in a Diabetic Surgical Population Versus a Non-diabetic Surgical Population.
Brief Title: Residual Gastric Volume Measured by Ultrasound in Diabetic Surgical Population Versus Non-diabetic Surgical Population.
Status: Completed | Type: Observational
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Responsible Party: Principal Investigator, Jose Alfonso Sastre, Principal Investigator, Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León
Other Study IDs: PI 2022 02 934
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Gastric ultrasound; Full stomach; Surgery
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Diabetic patients: Diabetic patients undergoing scheduled surgery
- Non-diabetic patients: Non-diabetic patients undergoing sheduled surgery

SUMMARY:
Comparison of residual gastric volume measure by ultrasounds between diabetic and non-diabetic patients scheduled for elective surgery

DETAILED DESCRIPTION:
The presence of gastric content increases the risk of aspiration during general anesthesia. Delayed gastric emptying has been described in diabetic patients; for that reason, diabetic patients could have a high risk of aspiration despite adequate fasting. This study aimed to compare ultrasound-guided measurement of residual gastric volume between diabetic and non-diabetic patients scheduled for elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI<40 kg.m-2;
* Age over 18 years;
* American Society of Anesthesiologists' physical status status I-III
* who were to undergo elective surgery and had the ability to understand the rationale of the study and provide informed consent

Exclusion Criteria:

* Pregnancy
* Recent upper gastrointestinal bleed (< 1 month)
* Abnormal anatomy of the upper gastrointestinal tract (such as hiatal hernias and gastric tumors)
* Previous surgical procedures on the esophagus, stomach, or upper abdomen
* Gastroesophageal reflux disease
* Previous use of prokinetics or high doses of opiates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fasted diabetic and non-diabetic patients scheduled for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Residual gastric volume | Preoperative
  Residual gastric volume measured by ultrasounds

SECONDARY OUTCOMES:
Antral cross-sectional area | Preoperative
  Antral cross-sectional area measured by ultrasounds

CONTACTS AND LOCATIONS:
Overall Officials: José A. Sastre, MD, PhD, Principal Investigator — Anesthesiology Service. Salamanca University Hospital
Locations (1):
- IBSAL, Salamanca, Salamanca, Spain

REFERENCES:
- [Background] Sastre JA, Lopez T, Julian R, Bustos D, Sanchis-Dux R, Molero-Diez YB, Sanchez-Tabernero A, Ruiz-Simon FA, Sanchez-Hernandez MV, Gomez-Rios MA. Assessing Full Stomach Prevalence with Ultrasound Following Preoperative Fasting in Diabetic Patients with Dysautonomia: A Comparative Observational Study. Anesth Analg. 2024 Dec 1;139(6):1300-1308. doi: 10.1213/ANE.0000000000007110. Epub 2024 Aug 8. PMID 39116006